CLINICAL TRIAL: NCT01208779
Title: An Epidemiological, Non-interventional Study to Evaluate Patient Compliance in Postmenopausal Women With Estrogen Receptor Positive Breast Cancer
Brief Title: Epidemiology Study in Postmenopausal Women With Estrogen Receptor Positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ORS-DUM-2010/1
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Hormon Receptor Positive Breast Cancer
Keywords: Compliance; HR+ breast cancer; epidemiology
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women with estrogen receptor positive breast cancer already receiving treatment with an aromatase inhibitor (AI) will be enrolled in the study

SUMMARY:
This observational study in estrogen receptor positive early breast cancer patients is aimed to evaluate the patients' compliance to aromatase inhibitor (AI) therapy and to collect country-specific data in estrogen receptor positive early breast cancer patients including data on demography, disease characteristics and disease management.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females with estrogen receptor positive breast cancer that are currently treated with aromatase inhibitor (AI) medication
* Provision of subject informed consent

Exclusion Criteria:

* If participating in any clinical trial, the subject cannot take part in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncology centers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Evaluate compliance rate, as assessed by investigator, after 12 months from baseline. | 12 months

SECONDARY OUTCOMES:
Evaluate compliance rate, assessed by investigator, after 6 months of follow up | 12 months
Evaluate the extent of patient educational activities as assessed by patient (using patient questionnaire) after 6 and 12 months | 12 months
Evaluate patient compliance as assessed by the patient (using patient questionnaire) after 6 and 12 months | 12 months
Collect epidemiology data; Demographic data: age, height, weight, lifestyle, menarche, childbirth, lactation, menopausal status | 12 months
Primary disease (breast cancer) characteristics: receptor status, disease stage | 12 months
Disease management data: treatment/treatment changes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jasna Pesic, Principal Investigator — M.D.spec of oncology, Institute for oncology Vojvodina, Sremska Kamenica
Locations (2):
- Serbia (2):
  - Research Site, Vojvodina, Sremska Kamenica
  - Research Site, Belgrade